CLINICAL TRIAL: NCT01968928
Title: The Role of Pyruvate Kinase M2 in Growth, Invasion and Drug Resistance in Human Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201308044RIN
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Bladder Urothelial Carcinoma
Keywords: Bladder urothelial carcinoma (UC); pyruvate kinase; drug resistance; shikonin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: None Retained — Tissue samples of tumors as well as normal-appearing mucosa collected in the tissue bank are to be used to examine the cellular and molecular events involved. Comparisons will be made to differentiate cellular changes between tumors and the normal counterparts.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- drug-resistant: specimens com from drug-resistant bladder urothelial carcinoma patients.
- normal: specimens come from normal bladder urothelial carcinoma patients.
- non-tumoral: specimens come from non-tumoral patients.

SUMMARY:
Bladder urothelial carcinoma (UC) is a common malignancy and the incidence is increasing by years in Taiwan. Chemoresistance was inevitable in treatment of metastatic disease and lead to the ominous outcomes. To develop novel therapeutic strategies to overcome chemoresistance is imperative. Cancer cells uptake glucose at higher rates than normal tissue but use most of glucose for glycolysis even under normoxia condition, which is known as the Warburg effect. Pyruvate kinase (PK) catalyzes the last step in the process of glycolysis, and one of it isoform--PKM2 has been reported to be associated with tumor progression and some specific tissues and promotes the Warburg effect in cancer cells.

DETAILED DESCRIPTION:
Regulation of PKM2 can be a novel target of cancer therapy. Meanwhile, PKM2 may play a critical role in the development of drug resistance and can be a promising target to overcome drug resistance.

In this study, our specific aims are as follows:

1. To prove the differentia expression levels of PKM2 in UC cells and drug-resistant UC cells, as well as in human UC tissues and drug-resistant UC tissues.
2. To examine the effect of PKM2 regulations（PKM2 siRNA and shikonin）on invasiveness and metastatic ability of UC cells and clarify the role of PKM2 in human UC cells.
3. To investigate the combinatory effect of PKM2 regulations（PKM2 siRNA and shikonin）and currently used chemotherapeutic agents (cisplatin，gemcitabine ,doxorubicin). Do PKM2 regulations enhance the cytotoxic effect of chemotherapy and overcome the chemoresistance？
4. To further prove the in vitro findings in the nude mice xenograft model。

ELIGIBILITY:
Inclusion Criteria:

* patients with age between 20-80 years old and had taken Radical Cystectomy or nephrectomy between 2008-2012

Exclusion Criteria:

* patients with age not located in the interval of 20-80 years old.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with age between 20-80 years old and had taken Radical Cystectomy or nephrectomy between 2008-2012 were chosen as study population.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The IHC score | at the time of surgery
  the IHC scores are acquired by IHC staining and the comparisons between each specimen are determined by IHC scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-How Huang, M.D., Ph.D., Principal Investigator — Department of Urology, National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- Department of Urology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Vander Heiden MG, Cantley LC, Thompson CB. Understanding the Warburg effect: the metabolic requirements of cell proliferation. Science. 2009 May 22;324(5930):1029-33. doi: 10.1126/science.1160809. PMID 19460998
- [Background] Christofk HR, Vander Heiden MG, Harris MH, Ramanathan A, Gerszten RE, Wei R, Fleming MD, Schreiber SL, Cantley LC. The M2 splice isoform of pyruvate kinase is important for cancer metabolism and tumour growth. Nature. 2008 Mar 13;452(7184):230-3. doi: 10.1038/nature06734. PMID 18337823
- [Background] Chen J, Xie J, Jiang Z, Wang B, Wang Y, Hu X. Shikonin and its analogs inhibit cancer cell glycolysis by targeting tumor pyruvate kinase-M2. Oncogene. 2011 Oct 20;30(42):4297-306. doi: 10.1038/onc.2011.137. Epub 2011 Apr 25. PMID 21516121
- [Background] Yang W, Lu Z. Regulation and function of pyruvate kinase M2 in cancer. Cancer Lett. 2013 Oct 10;339(2):153-8. doi: 10.1016/j.canlet.2013.06.008. Epub 2013 Jun 18. PMID 23791887